CLINICAL TRIAL: NCT05995717
Title: An Acceptability Study to Evaluate the Compliance, Gastrointestinal Tolerance, Palatability and Metabolic Control of Children With Phenylketonuria (PKU) When Using PKU UP (a Food for Special Medical Purposes) as Part of Dietary Management.
Brief Title: Evaluation of PKU UP
Acronym: PKU UP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Collaborators: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-PAED-LIQ-2022-10-07; 327641 (Other: IRAS); 23/NW/0185 (Other: UK REC - North West Liverpool Central)
Record Dates: First submitted 2023-08-03; First posted 2023-08-16 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: PKU
Keywords: Phenylketonuria; PKU; Glyco-Macro-Peptide; GMP; amino acid; AA; protein substitute; PS; United Kingdom; UK; children; PKU UP; Glycomacropeptide
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PKU UP (Experimental): All participants will be assessed by their dietitian and prescribed an appropriate amount of the study product, PKU UP, to manage their phenylketonuria.
  Interventions: Dietary Supplement: PKU UP

INTERVENTIONS:
Dietary Supplement: PKU UP — PKU UP is a food for special medical purposes (FSMP). This product is for use in the dietary management of Phenylketonuria (PKU) in children aged from one (1) to ten (10) years.
  PKU UP is a neutral-flavoured, ready-to-drink, low-phenylalanine protein substitute containing a blend of glycomacropeptide (GMP) isolate, essential and non-essential amino acids, fat, carbohydrate, vitamins, minerals and docosahexaenoic acid (DHA).

SUMMARY:
PKU UP is a prospective, single-arm, open-label, 26-week acceptability study to evaluate PKU UP for the dietary management of participants with phenylketonuria (PKU). Up to 15 participants aged 1 - 10 years old will be recruited and it is anticipated the study will open in at least three sites in the United Kingdom (UK) to recruit the target number of participants in the required timeframe.

DETAILED DESCRIPTION:
PKU is a rare inborn error of metabolism with a prevalence of 1 in 10,000 in the UK population. The mainstay of treatment for most individuals is dietary therapy with a strict protein-restricted diet. We propose to recruit children with a diagnosis of PKU aged 1-10 years.

The study product, PKU UP, is a food for special medical purposes (FSMP), as defined by the Delegated Act EU 2016/128, used for the dietary management of Phenylketonuria (PKU).

The study will be investigating the acceptability of PKU UP, as defined by the Advisory Committee on Borderline Substances (ACBS). This includes the following:

* participant adherence to recommended intakes
* gastrointestinal symptoms
* evaluations of palatability.

Each participant will be on the study for 26 weeks. This includes evaluation part 1 and evaluation part 2:

* Part 1 consists of a 12 week period where participants introduce the study product into their diet. Gastrointestinal tolerance, metabolic control, compliance, product acceptability and dietary quality will be evaluated.
* Part 2 consists of a 14 week period where participants continue to take the study product for a longer assessment of growth and nutritional status.

Data collection will be performed using paper and/or electronic Case Report Forms completed by the investigators at the baseline, evaluation periods and end of study visits. There will also be three questionnaires completed by the parents/guardians over the course of the study, in relation to protein substitute intake, gastrointestinal tolerance, and product acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU requiring a low-protein diet and protein substitute.
* Participants who are adherent with their blood phenylalanine (Phe) testing, in the opinion of the investigator.
* Participants aged 1-10 years.
* Participants who in the opinion of the investigator are anticipated to be able to take at least half of their daily protein equivalent requirement from PKU UP (in order to assess this, a taste test (or similar) may be conducted at investigator's discretion as part of the screening process).
* Willingly given, written, informed consent from the parent(s)/guardian(s).
* Willingly given, written assent by the participant (if appropriate).

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator.
* Any co-morbidity, which, in the opinion of the investigator, would preclude participation in the study.
* Diagnosis of persistent hyperphenylalaninemia, or mild PKU not requiring a low protein diet and protein substitute.
* Allergy or intolerance to milk.
* Participants who are currently participating in, plan to participate in or have participated in an interventional investigational drug, food or medical device study within 30 days prior to the screening visit.
* Use of additional micronutrient supplements during the evaluation period, unless clinically indicated and prescribed by the Investigator (must be recorded in both the medical records and case report form).

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in phe level between baseline and visit 3 | 26 weeks
  Change in phe level as measured by dried blood spot testing
Change in tyrosine level between baseline and visit 3 | 26 weeks
  Change in tyrosine level as measured by dried blood spot testing
Change in PI impression of metabolic control | Week 0, week 6, week 12, week 26
  Assessment of the participant's metabolic control in the opinion of the investigator
Change in the growth of participants as measured by Height (length in under 2 years of age), Head circumference in under 2 years of age and Weight. | Week 0, week 12, week 26
  Assessed via anthropometry measurements. Participants will be weighed and measured for growth monitoring.
Change in GI tolerance (participant) | Week 0, week 6, week 12, week 26
  Gastrointestinal tolerance assessed using the PedsQL Gastrointestinal Symptoms Scale completed by the participants
Change in PI impression of GI tolerance | Week 0, week 6, week 12, week 26
  Assessment of the participant's GI tolerance in the opinion of the investigator
Change in compliance with study product consumption | Week 0, week 6, week 12, week 26
  Assessed via participant diary regarding study product intake
Change in PI impression of study product intake | Week 0, week 6, week 12, week 26
  Assessment of the participant's compliance in the opinion of the investigator
Change in product acceptability | Week 0, week 12, week 26
  Assessed via a product acceptability questionnaire completed by the participant/parent
Change in dietary intake | Week 0, week 12, week 26
  Assessed via 24-hour recall and low protein food frequency questionnaire
Change in nutritional biochemistry | Week 0, week 26
  Assessed via venous blood sample of approximately 10ml

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Children's Hospital, Birmingham
  - St. Luke's Hospital, Bradford
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Nottingham Children's Hospital, Nottingham
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No